CLINICAL TRIAL: NCT00678795
Title: A Double Blind, Randomised, Placebo Controlled, Parallel Group Study of Cannabis Based Medicine (CBM) Extract, in Patients Suffering Detrusor Overactivity Associated With Multiple Sclerosis.
Brief Title: A Parallel Group Study to Compare Sativex® With Placebo in the Treatment of Detrusor Overactivity in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWMS0208
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Detrusor Overactivity; Multiple Sclerosis
Keywords: Detrusor overactivity; Multiple Sclerosis
MeSH Terms: conditions — Urinary Bladder, Overactive; Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental): Each 100 ul actuation contains 27 mg delta-9-tetrahydrocannabinol (THC) and 25 mg cannabidiol (CBD). A maximum of 48 actuations (130 mg of THC and 120 mg of CBD) was permitted in any 24 hour period.
  Interventions: Drug: Sativex®
- Placebo (Placebo Comparator): Each 100 ul actuation contains the colorants plus excipients. A maximum of 48 actuations was permitted in any 24 hour period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex® — Containing ∆9 tetrahydrocannabinol (THC), 27 mg/ml and cannabidiol (CBD), 25 mg/ml as extract of Cannabis sativa L.
  Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three-hour period and 48 actuations (THC 130 mg:CBD 120 mg) in 24 hours
  Other Names: GW-10000-02
  Arms: Sativex
Drug: Placebo — containing excipients only. Subjects received study medication delivered in 100 µl actuations from a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three-hour period and 48 actuations in 24 hours.
  Other Names: GW-4001-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Sativex® compared with placebo in reducing the daily number of episodes on incontinence.

DETAILED DESCRIPTION:
This is a ten week, multicentre, double blind, randomised, placebo controlled parallel group study to evaluate the efficacy of Sativex® on urge incontinence associated with neurogenic unstable bladder. Multiple sclerosis patients with incontinence symptoms are screened to determine eligibility and complete a two-week baseline period. They then return for a further eligibility check, randomisation and initial dosing. Subjects titrate and self-medicate with study medication between study visits at weeks two and five. They will also complete efficacy assessments in their diary-books and at visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female, aged 18 years or over.
* Diagnosed with MS and with detrusor overactivity not wholly relieved by current therapy.
* At least three incontinence episodes within five consecutive days during the baseline period
* Stable dose of anticholinergic medication for at least 14 days leading to study entry.
* Agreement, if female and of child bearing potential or if male with a partner of child bearing potential, to ensure that effective contraception is used during the study and for three months thereafter.
* Has not used cannabinoids (including cannabis, Marinol® or nabilone) for at least seven days before Visit 1 and willing to abstain from any use of cannabinoids during the study.
* Agreement for the UK Home Office, their general practitioner, and their consultant if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* A symptomatic UTI or any cause of detrusor overactivity other than neurogenic causes due to MS.
* Using ISC.
* A history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* A history of alcohol or substance abuse.
* A severe cardiovascular disorder, such as ischaemic heart disease, arrhythmias (other than well controlled atrial fibrillation), poorly controlled hypertension or severe heart failure.
* A history of epilepsy.
* If female, are pregnant of lactating, or are planning a pregnancy to occur during the course of the study.
* Significant renal or hepatic impairment.
* Elective surgery or other procedures requiring general anesthesia scheduled to occur during the study.
* Terminal illness or any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or influence the result of the study, or the subjects ability to participate in the study.
* Regular levodopa (Sinement®, Sinement Plus®, Levodopa, L-dopa, Madopar®, Benserazide) within the seven days leading up to study entry.
* Receiving and unwilling to stop fentanyl for the duration of the study.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medications.
* Intention to travel internationally or to donate blood during the study.
* Participation in another research study in the 12 weeks leading up to study entry.
* Previous randomization in to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2002-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cris Constantinescu, MD PhD, Principal Investigator — Division of Clinical Neurology, Queen's Medical Centre
Locations (1):
- Division of Clinical Neurology, Queen's Medical Centre, Nottingham, Notts, United Kingdom

REFERENCES:
- [Result] Kavia RB, De Ridder D, Constantinescu CS, Stott CG, Fowler CJ. Randomized controlled trial of Sativex to treat detrusor overactivity in multiple sclerosis. Mult Scler. 2010 Nov;16(11):1349-59. doi: 10.1177/1352458510378020. Epub 2010 Sep 9. PMID 20829244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 67 | 68
Completed | 56 | 62
Not Completed | 11 | 6
Not completed — Adverse Event | 7 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 66 | 129
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.61 (9.31) | 46.79 (11.20) | 47.69 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 98
  Male | 15 | 22 | 37
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35 | 33 | 68
  Belgium | 23 | 26 | 49
  Romania | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Daily Number of Incontinence Episodes at the End of Treatment
Description: To assess the effect of Sativex in neurogenic overactive bladder, the incontinence episode frequency was selected as the primary endpoint. Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 10 weeks
Population: All randomised subjects who received at least one dose of study medication and had on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of daily episodes
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 60 | 64
number of daily episodes | -1.08 (1.42) | -0.99 (1.09)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The primary endpoint, the change in the number of incontinence episodes per day, was compared between treatment groups using analysis of covariance (ANCOVA). The model included treatment and centre as factors and baseline number of incontinence episodes per day as a covariate; Test type: Superiority or Other; p = 0.569, ANCOVA; Estimated mean treatment difference = -0.11, 95% CI 2-sided [-0.47 to 0.26]

2. Secondary Outcome: Change From Baseline in the Mean Daily Episodes of Urgency at the End of Treatment
Description: Subjects documented in the daily subject diary each instance of urgency, and the time that each took place, as for the recording of incontinence episode frequency. Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: Daily diary entries throughout 10 week study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of daily episodes
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 60 | 64
number of daily episodes | -1.91 (2.44) | -1.12 (2.80)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the number of urgency episodes per day was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline number of urgency episodes per day as a covariate; Test type: Superiority or Other; p = 0.071, ANCOVA; Estimated mean treatment difference = -0.76, 95% CI 2-sided [-1.58 to 0.07]

3. Secondary Outcome: Change From Baseline in the Mean Daily Episodes of Nocturia at the End of Treatment
Description: Subjects documented in the daily subject diary each instance of nocturia, and the time that each took place (as for the recording of incontinence episode frequency). Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of daily episodes
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 60 | 64
number of daily episodes | -0.55 (0.75) | -0.21 (0.70)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the number of nocturia episodes per day was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline number of nocturia episodes per day as a covariate; Test type: Superiority or Other; p = 0.010, ANCOVA; Estimated mean treatment difference = -0.28, 95% CI 2-sided [-0.50 to -0.07]

4. Secondary Outcome: Change From Baseline in the Mean Daily Number of Incontinence Pads Used at the End of Treatment
Description: Subjects documented in the daily subject diary, the total number of incontinence pads they had used each day. Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pads used daily
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 48 | 55
pads used daily | -0.88 (1.50) | -0.73 (1.64)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the number of incontinence pads used per day was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline number of number of incontinence pads used per day as a covariate; Test type: Superiority or Other; p = 0.74, ANCOVA; Estimated mean treatment difference = -0.08, 95% CI 2-sided [-0.57 to 0.41]

5. Secondary Outcome: Change From Baseline in Mean Total Incontinence Quality of Life (I-QOL) Questionnaire Score at the End of Treatment (Completion or Withdrawal)
Description: The I-QOL consists of 22 items from three subscales; avoidance/limiting behaviour (eight items), psychosocial impact (nine items) and social embarrassment (five items). The responses to each of the 22 items were summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation. The transformation formula used for the I-QOL total scores is: Transformed score = 100 x (the sum of the items - lowest possible score) / Possible raw score range. An increase in score indicates an improvement in QOL.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 59 | 61
units on a scale | 14.21 (17.51) | 9.58 (12.77)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in the I-QOL score at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline I-QOL score as a covariate; Test type: Superiority or Other; p = 0.166, ANCOVA; Estimated mean treatment difference = 3.90, 95% CI 2-sided [-1.65 to 9.46]

6. Secondary Outcome: Change From Baseline in Mean Overall Bladder Condition 0-10 Numerical Rating Scale Score at the End of Treatment
Description: Subjects subjectively assessed the severity of their urinary incontinence and general bladder symptoms by responding to the following question on a Numerical Rating Scale: My bladder condition, taking everything into account, causes me: 0 = "no problems" and 10 = "intolerable problems". Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 61 | 66
units on a scale | -2.3 (2.16) | -0.9 (2.04)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in the overall bladder condition Numerical Rating Scale score at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline overall bladder condition Numerical Rating Scale score as a covariate; Test type: Superiority or Other; p = 0.001, ANCOVA; Slope = -1.16, 95% CI 2-sided [-1.82 to -0.51]

7. Secondary Outcome: Patient's Global Impression of Change
Description: Subjects were asked at completion or withdrawal to give their impression of the overall change in their condition since entry into the study using the following seven-point scale: 1 = 'Very Much Improved', 2 = 'Much Improved', 3 = 'Minimally Improved', 4 = 'No Change', 5 = 'Minimally Worse', 6 = 'Much Worse', 7 = 'Very Much Worse'. The numbers who scored 1, 2, or 3 are presented.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 63 | 67
participants | 51 | 39
Statistical Analysis 1: Comparison: Sativex vs Placebo; For Patient Global Impression of Change, the proportions of subjects who considered their condition 'Very Much Improved', 'Much Improved' or 'Minimally Improved' were compared between treatment groups using Fisher's Exact Test; Test type: Superiority or Other; p = 0.002, Fisher Exact; Estimated mean treatment difference = 25.40, 95% CI 2-sided [10.37 to 40.42]

8. Secondary Outcome: Change From Baseline in the Mean Number of Daily Voids at the End of Treatment
Description: Baseline was the average of all available data recorded during the 14 days immediately prior to the randomisation visit. End of Treatment was the last average available from Week 3, Week 5, and Weeks 7-8. A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of daily episodes
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 60 | 64
number of daily episodes | -1.73 (1.95) | -0.87 (1.86)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the number of voids per day was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline number of voids per day as a covariate; Test type: Superiority or Other; p = 0.007, ANCOVA; Estimated mean treatment difference = -0.85, 95% CI 2-sided [-1.47 to -0.23]

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the extension study onset to the last study visit (up to 99 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 2/67 | 2/68
Other Adverse Events (participants affected / at risk) | 48/67 | 43/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=67) | Placebo (N=68)
Vomiting (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=67) | Placebo (N=68)
Vomiting Not Otherwise Specified (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Diarrhoea Not Otherwise Specified (Gastrointestinal disorders) | 2 | 4
Feeling Drunk (General disorders) | 3 | 0
Weakness (General disorders) | 3 | 2
Fatigue (General disorders) | 0 | 3
Application Site Pain (General disorders) | 0 | 3
Urinary tract infection Not Otherwise Specified (Infections and infestations) | 4 | 7
Cystitis Not Otherwise Specified (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Dizziness (Nervous system disorders) | 12 | 5
Headache Not Otherwise Specified (Nervous system disorders) | 5 | 5
Balance Impaired Not Otherwise Specified (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 3
Disorientation (Psychiatric disorders) | 4 | 0
Dissociation (Psychiatric disorders) | 4 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Feeling Abnormal (General disorders) | 2 | 0
Chest Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Influenza (Infections and infestations) | 0 | 2
Pharyngitis Viral Not Otherwise Specified (Infections and infestations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Disturbance in Attention (Nervous system disorders) | 2 | 0
Memory Impairment (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 2
Confusion (Psychiatric disorders) | 2 | 0
Sweating Increased (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.